CLINICAL TRIAL: NCT01078194
Title: Observational Study on the Secondary Placement of the A.M.I. Soft Gastric Band in Weight Regain or Weight Loss Failure After Lap. Gastric Bypass
Brief Title: Secondary Bypass Banding for Weight Regain or Weight Loss Failure After Lap. Gastric Bypass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gerhard Prager / M.D., Medical University of Vienna / Department of Surgery
Other Study IDs: MUW ADIP STUDY 16
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-01

CONDITIONS: Morbid Obesity
Keywords: Weight regain; Weight loss failure; Gastric bypass
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Weight regain / weight loss failure: Weight regain of more than 10 kg from or weight loss of less than 50% EWL 18 months after lap. gastric bypass
  Interventions: Device: Secondary Bypass Banding (adjustable A.M.I. Soft Gastric Band)

INTERVENTIONS:
Device: Secondary Bypass Banding (adjustable A.M.I. Soft Gastric Band) — Secondary Placement of the A.M.I. Soft Gastric Band for laparoscopic bypass banding
  Other Names: A.M.I. Soft Gastric Band

SUMMARY:
This is an observational study on the efficacy of the secondary placement of the A.M.I Soft Gastric Band in weight regain or weight loss failure after lap. gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Weight regain of more than 10 kg from nadir
* Excessive weight loss of less than 50% at 18 months after laparoscopic gastric bypass

Exclusion Criteria:

* Formerly leak at the gastrojejunostomy
* Formerly open abdominal surgery
* Anastomotic ulcer

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Weight regain of more than 10 kg from nadir or weight loss failure defined as excessive weight loss of less than 50% 18 months after laparoscopic gastric bypass
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 2 years
  Excessive weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Prager, M.D., Principal Investigator — Medical University of Vienna, Department of Surgery
Locations (1):
- Medical University of Vienna, Department of Surgery, Vienna, Austria